CLINICAL TRIAL: NCT06391073
Title: Reach Out 2: Randomized Clinical Trial of Emergency Department-Initiated Hypertension Mobile Health Intervention Connecting Multiple Health Systems
Brief Title: Reach Out 2: Emergency Department-Initiated Hypertension Mobile Health Intervention Connecting Multiple Health Systems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Michigan (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Lesli Skolarus, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MD019124 (NIH)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): The usual care group is standard of care. They will receive the standard ED discharge materials available as recommended by their ED physician. These materials recommend lifestyle changes, dietary changes, medication as directed, and follow-up with a PCP as directed.
- REACH OUT (Experimental): REACH OUT messaging is based on BP control. Control is defined as SMBP <135/85. Every 4 weeks SMBP measurements will be assessed and mHealth components will be escalated, de-escalated, or remain the same.
  If BP is controlled, SMBP prompts will be sent once a week and there will be no facilitated appointments.
  If BP is uncontrolled, SMBP prompts will be sent three times per week and facilitated provider scheduling and transportation will occur.
  Participants will have the option include a partner, friend, or family member with text-messaging capability who could support them on their BP journey. The partner will receive Reach Out materials and text messages to remind the participant to engage in SMBP and of their upcoming appointments (if uncontrolled).
  Interventions: Behavioral: Self-Measured Blood Pressure Monitoring; Behavioral: Physician appointment and transportation scheduling

INTERVENTIONS:
Behavioral: Self-Measured Blood Pressure Monitoring — Prompted SMBP with tailored feedback
  Arms: REACH OUT
Behavioral: Physician appointment and transportation scheduling — Physician appointment and transportation scheduling or none dependent on current BP control
  Arms: REACH OUT

SUMMARY:
Emergency department visits provide an opportunity to identify people with undiagnosed, untreated, or uncontrolled high blood pressure. In Reach Out, we will test whether a mobile health intervention yields a greater reduction in blood pressure than usual care among individuals identified with high blood pressure during a safety-net emergency department visit. Subsequently, we will estimate the reduction in heart attack, stroke, and dementia if Reach Out were implemented across all U.S. safety-net emergency departments.

DETAILED DESCRIPTION:
Hypertension is the most important modifiable risk factor for cardiovascular disease. Black Americans have the highest prevalence of hypertension and the lowest rates of blood pressure (BP) control of any racial or ethnic group in the U.S., contributing to cardiovascular disease disparities. Low-income Americans are also disproportionally burdened by hypertension. To achieve health equity, new approaches to hypertension management leveraging safety-net healthcare systems to reach underserved populations are needed.

One approach to addressing the hypertension epidemic is to identify and treat people undiagnosed, untreated, or with undertreated hypertension - people who have fallen through the cracks in the healthcare system. We did this in Reach Out 1 (R01MD011516), a mobile health (mHealth) 8-arm factorial trial of hypertensive patients recruited from a safety-net ED. Overall, systolic BP declined by 9.2 mmHg (95% CI -12.2 to - 6.3) after 6 months, without differences across treatment arms. Reach Out 1 successfully enrolled a hypertensive, medically underserved population into a mHealth intervention. Despite a very large reduction in BP overall, the efficacy of the Reach Out mHealth intervention is uncertain, given the lack of a control group.

Reach Out 2 proposes to test the most promising components of Reach Out 1 in a randomized open, blinded-endpoint (PROBE) controlled trial. Reach Out 2, continues our work with the same safety-net ED and Federally Qualified Health Centers. In Reach Out 2, we will compare usual care, to 6-months of prompted self-monitored blood pressure (SMBP) monitoring with tailored feedback and facilitated primary care appointment and transportation. The usual care group will receive instructions to follow up with a primary care provider after ED discharge. After 6 months, the intervention participants will enter an extended treatment period of long-term SMBP monitoring. To contextualize our findings, we will use our chronic disease agent-based simulation model to estimate the reduction in myocardial infarction, stroke, and dementia if Reach Out 2 were to be implemented in safety-net EDs across the US. The overarching goal of our proposal is to determine whether a low-tech mHealth intervention will reduce BP more than usual care among patients recruited from a safety-net ED and to understand the potential national impact of such an intervention. Because safety-net EDs are anchor institutions that care for large populations of medically underserved hypertensive people, mHealth strategies initiated here have tremendous potential to reduce cardiovascular inequities. To reach this potential, evidence based interventions to reduce BP must be identified (aim 1), long-term engagement evaluated (aim 2), and their impact understood (aim 3).

ELIGIBILITY:
While in the ED, the patient must meet all of the following:

* Adult (≥18 y/o)
* At least one BP with Systolic BP ≥160 or a Diastolic BP ≥100 (criteria 1)
* If the patient has repeated measurements after achieving Criteria 1, at least one of the repeat BP remains systolic BP ≥140 or a diastolic BP ≥90
* Must have cell phones with text-messaging capability
* Likely to be discharged from the ED

Exclusion Criteria for Main Trial Participants:

* Critical illness
* Unable to read English (<1% at study site)
* Incarcerated
* Pregnant
* Pre-existing condition making 6-month follow-up unlikely

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 6 month
  Change in 6-month Systolic Blood Pressure (SBP)

SECONDARY OUTCOMES:
Change in diastolic blood pressure | 6 month
  Change in 6-month Diastolic Blood Pressure (DBP)
BP Control (130/80mmHg) | 6 month
  Proportion of participants with controlled BP at 6-months. BP control is defined as BP less than 130/80 mmHg.

OTHER OUTCOMES:
BP Control (140/90mmHg) | 6 month
  Proportion of participants with controlled BP at 6-months. BP control defined as BP less than 140/90
Initiation of antihypertensive medication | 6 month
Change in antihypertensive medication | 6 month
Establishment of primary care | 6 month
  Time from ED visit to arrival at first primary care visit
Participant adherence with self-measured blood pressure monitoring | 6 month
  Proportion of BPs received after a BP prompt

CONTACTS AND LOCATIONS:
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data in which direct and indirect identifiers have been removed will be made available through data-sharing website
Supporting Information: Study Protocol
Time Frame: Before completion of trial data collection.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT06391073/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT06391073/ICF_001.pdf